CLINICAL TRIAL: NCT05095454
Title: A Pilot Study to Compare Short-Term Transcutaneous or Epidural Spinal Stimulation for Enabling Motor Function in Humans With Spinal Cord Injury
Brief Title: Short-Term Transcutaneous or Epidural Spinal Stimulation for Enabling Motor Function in Humans With SCI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kristin Zhao, PhD (Other)
Responsible Party: Sponsor-Investigator, Kristin Zhao, PhD, Principal Investigator, Mayo Clinic
Organization: Mayo Clinic (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 21-006340
Record Dates: First submitted 2021-10-03; First posted 2021-10-27 (Actual); Results first posted 2024-07-09 (Actual); Last update posted 2024-07-09 (Actual); Status verified 2024-06

CONDITIONS: Paraplegia; Tetraplegia; Paralysis; Quadraplegia
MeSH Terms: conditions — Paraplegia; Quadriplegia; Paralysis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Percutaneous Epidural Stimulation (Experimental): Epidural spinal stimulation will be delivered via percutaneously implanted electrodes during rehabilitation. All implanted electrodes will be removed at the end of trial participation. The effects of epidural stimulation will be recorded via electrophysiological and biomechanical metrics described within the outcomes measures.
  Interventions: Device: Percutaneous epidural electrical spinal stimulation
- Transcutaneous Epidural Stimulation (Experimental): Transcutaneous spinal stimulation will be delivered via skin surface-level electrodes during rehabilitation. The effects of transcutaneous stimulation will be recorded via electrophysiological and biomechanical metrics described within the outcomes measures.
  Interventions: Device: Transcutaneous electrical spinal stimulation

INTERVENTIONS:
Device: Percutaneous epidural electrical spinal stimulation — Abbott percutaneous trial lead for epidural neurostimulation (Model 3086)
  Ripple Neuromed Nomad Neurostimulation System
  Arms: Percutaneous Epidural Stimulation
Device: Transcutaneous electrical spinal stimulation — Digitimer DS8R Bipolar Constant Current Stimulator
  Arms: Transcutaneous Epidural Stimulation

SUMMARY:
A study comparing short-term delivery of epidural spinal stimulation versus transcutaneous spinal stimulation.

DETAILED DESCRIPTION:
The purpose of this study is to compare spinal motor nerve response to electrical stimulation delivered directly to the epidural space, and delivered through the skin (transcutaneously), and to measure any changes in motor performance over the course of about 5 months, during and after using one of the two types of stimulation.

ELIGIBILITY:
Inclusion Criteria:

* Spinal cord injury due to trauma located at or above the tenth thoracic vertebrae (T10)
* American Spinal Injury Association grading scale of A-D (2 from each) below the level of SCI
* Intact spinal reflexes below the level of SCI
* At least 1-year post-SCI
* At least 22 years of age
* Willing to use medically acceptable methods of contraception, if female and of child-bearing potential

Exclusion Criteria:

* Currently a prison inmate, or awaiting trial, related to criminal activity
* Pregnancy at the time of enrollment
* History of chronic and/or treatment resistant urinary tract infection
* Unhealed decubitus ulcer
* Unhealed skeletal fracture
* Untreated clinical diagnosis of depression
* Undergoing, or planning to undergo, diathermy treatment
* Active participation in another interventional clinical trial
* Presence of conditions or disorders which require MRI monitoring
* A history of coagulopathy or other significant cardiac or medical risk factors for surgery
* Current use of a ventilator
* Clinically diagnosed cardiopulmonary complications such as chronic obstructive pulmonary disease, cardiac failure, or heart arrhythmia that contraindicate changes in body position such as supine-to-sit-to-stand activities, prolonged standing, or stepping
* History of frequent hypotension characterized by light headedness, or loss of consciousness
* History of frequent hypertension characterized by headache, or bradycardia
* History of frequent, severe, autonomic dysreflexia
* Any illness or condition which, based on the research team's assessment, will compromise with the patient's ability to comply with the protocol, patient safety, or the validity of the data collected during this study.

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2022-03-04 (Actual); Primary Completion 2023-03-30 (Actual); Study Completion 2023-03-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kristin D Zhao, Ph.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Veith DD, Gill ML, Beck LA, Whitmarsh CL, Fernandez KA, Linde MB, Asp AJ, Mills CJ, Bendel MA, Grahn PJ, Zhao KD. Functional outcomes and participants' perspectives during short-term application of spinal stimulation in individuals with spinal cord injury. J Spinal Cord Med. 2025 Nov;48(6):978-989. doi: 10.1080/10790268.2024.2383377. Epub 2024 Aug 22. PMID 39172032

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment was conducted from March 4, 2022 to October 11, 2022 within a medical clinic.
Groups:
- Percutaneous Epidural Stimulation: Epidural spinal stimulation will be delivered via percutaneously implanted electrodes during rehabilitation. All implanted electrodes will be removed at the end of trial participation. The effects of epidural stimulation will be recorded via electrophysiological and biomechanical metrics described within the outcomes measures.
  Percutaneous epidural electrical spinal stimulation: Abbott percutaneous trial lead for epidural neurostimulation (Model 3086)
  Ripple Neuromed Nomad Neurostimulation System
Period: Overall Study
Arm/Group | Percutaneous Epidural Stimulation | Transcutaneous Epidural Stimulation
Started | 3 | 3
Completed | 3 | 2
Not Completed | 0 | 1
Not completed — Lengthy COVID-19 infection interrupted intervention to an unsatisfactory degree. | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Percutaneous Epidural Stimulation | Transcutaneous Epidural Stimulation | Total
Number analyzed (Participants) | 3 | 3 | 6
Age, Customized [Count of Participants; unit: Participants]
  22-29 | 2 | 2 | 4
  30-39 | 0 | 1 | 1
  40-49 | 1 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 3 | 3 | 6
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 3 | 3 | 6
  White | 2 | 3 | 5
  Black or African American | 0 | 0 | 0
  Multiracial | 0 | 0 | 0
  Other | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Electromyography
Description: Change in voltage measurements in major muscle groups below the level of injury. Specifically, change in soleus root mean square voltage during standing with and without stimulation.
Time Frame: Through study completion; an average of 5 months.
Measure: Mean (Standard Deviation); unit: volts
Arm/Group | Percutaneous Epidural Stimulation | Transcutaneous Epidural Stimulation
Number analyzed (Participants) | 3 | 3
volts | 0.00017507 (0.04279603) | 0.00006740 (0.05917040)

2. Primary Outcome: Foot Pressure
Description: Change in measurements of foot pressure in kilograms through shoe-insole pressure sensors.
Time Frame: Beginning of intervention to end of intervention, an average of 17 days.
Population: Increase in the difference in total loading force when standing, between beginning and end of intervention (an average of 17 days), with and without stimulation
Measure: Mean (Standard Deviation); unit: percentage of loading force increase
Arm/Group | Percutaneous Epidural Stimulation | Transcutaneous Epidural Stimulation
Number analyzed (Participants) | 3 | 1
percentage of loading force increase
  Beginning of intervention | 6 (9) | 0 (0)
  End of intervention | 40 (34) | 0 (0)

3. Primary Outcome: Somatosensory Evoked Potentials
Description: Measurements of change in voltage in the conduction of electricity through the peripheral nerves, cervical and lumbosacral spinal cord, deep brain structures, and sensory cortex, using surface electrodes.
Time Frame: Assessed at Baseline, 4 Weeks, 8 Weeks, and 20 Weeks; change from Baseline at week 20 reported.
Population: Change in amplitude of lumbar SSEP during tibial stimulation
Measure: Mean (Standard Deviation); unit: microvolts
Arm/Group | Percutaneous Epidural Stimulation | Transcutaneous Epidural Stimulation
Number analyzed (Participants) | 3 | 2
microvolts
  Left sided measurements | 0.67 (0.6) | 0.8 (0.99)
  Right sided measurements | 0.33 (0.12) | 0.35 (0.07)

4. Primary Outcome: Transcranial Magnetic Stimulation Motor Evoked Potentials
Description: Measurement of the threshold percentage change in voltage between pre-intervention and post-intervention in the first trapezius or deltoid muscle activated.
Time Frame: Assessed at Baseline, 4 Weeks, 8 Weeks, and 20 Weeks; change from Baseline at week 20 reported.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Percutaneous Epidural Stimulation | Transcutaneous Epidural Stimulation
Number analyzed (Participants) | 3 | 2
percent change | 3.33 (5.77) | 5 (7.07)

5. Primary Outcome: Injury Severity: International Standards for Neurological Classification of Spinal Cord Injury
Description: Change sensory and motor function impairment using the American Spinal Injury Association Impairment Scale. Individuals are classified from A" (complete SCI) to "E" (normal function). 28 dermatomes and 10 key muscles are assessed bilaterally. Summed results produce overall sensory and motor scores and combine with evaluation of anal sensory and motor function in determination of AIS classification. Sensory scores are rated 0 (sensation absent) to 2 (normal), bilaterally for each of 28 dermatomes. Muscle function is rated 0 (total paralysis) to 5 (active movement, full range of motion against significant resistance) for each myotome. Upper Extremity Motor Subscores and Lower Extremity Motor Subscores are scored from 0 to 50; the ASIA Motor Score is scored from 0 to 100. The presence of deep anal pressure and voluntary anal contraction are assessed as a yes/no; absence of these, in addition to sensory scores of 0 at S4-5 indicate a Complete injury (otherwise, the injury is Incomplete).
Time Frame: Assessed at Baseline, 4 Weeks, 8 Weeks, and 20 Weeks; change from Baseline at week 20 reported.
Measure: Number; unit: Participants
Arm/Group | Percutaneous Epidural Stimulation | Transcutaneous Epidural Stimulation
Number analyzed (Participants) | 3 | 2
Participants
  Change between Complete (C) and Incomplete (I) designations | 0 | 0
  Change in ASIA Impairment Scale (AIS) rating | 0 | 0
  Change in sensation of Deep Anal Pressure (DAP) | 0 | 0
  Change in Voluntary Anal Contraction (VAC) | 0 | 0

6. Primary Outcome: Patient-reported Bowel Function
Description: Measurement of change in bowel function using the Neurogenic Bowel Dysfunction Score. Answers to qualitative questions are rated from 0 to 5, with a higher number indicating more problematic symptoms, and totaled for a score which categorizes severity of neurogenic bowel symptoms. The total score ranges between 0 and 44 points. A higher total score indicates more severe bowel symptoms.
Time Frame: Assessed at Baseline, 4 Weeks, 8 Weeks, and 20 Weeks; change from Baseline at week 20 reported.
Measure: Mean (Full Range); unit: Score on a scale
Arm/Group | Percutaneous Epidural Stimulation | Transcutaneous Epidural Stimulation
Number analyzed (Participants) | 3 | 2
Score on a scale | -4 [-6 to -2] | -3.5 [-12 to 5]

7. Primary Outcome: Patient-reported Bladder Function
Description: Measurement of change in bladder function using the Neurogenic Bladder Symptom Score. Answers to qualitative questions are rated from 0 to 5, with a higher number indicating more problematic symptoms, and totaled for a score which categorizes severity of neurogenic bladder symptoms. The total score can range from 0 (no symptoms at all) to 74 (maximum symptoms).
Time Frame: Assessed at Baseline, 4 Weeks, 8 Weeks, and 20 Weeks; change from Baseline at week 20 reported.
Measure: Mean (Full Range); unit: Score on a scale
Arm/Group | Percutaneous Epidural Stimulation | Transcutaneous Epidural Stimulation
Number analyzed (Participants) | 3 | 2
Score on a scale | -11.3 [-12 to -8] | -4.5 [-6 to -3]

8. Primary Outcome: Male Patient-reported Sexual Function (1)
Description: Measurement of change in erectile dysfunction using the Sexual Health Inventory for Men (SHIM). Answers to qualitative questions are rated from 0 to 5, with a higher number indicating better erectile function, and totaled for a score which categorizes severity of erectile dysfunction. Total score can range from 1 to 25, with a lower number indicating more severe erectile dysfunction.
Time Frame: Assessed at Baseline, 4 Weeks, 8 Weeks, and 20 Weeks; change from Baseline at week 20 reported.
Measure: Mean (Full Range); unit: Score on a scale
Arm/Group | Percutaneous Epidural Stimulation | Transcutaneous Epidural Stimulation
Number analyzed (Participants) | 3 | 2
Score on a scale | -6.3 [-14 to 2] | 0 [-1 to 1]

9. Primary Outcome: Male Patient-reported Sexual Function (2)
Description: Measurement of change in erectile dysfunction using the International Index for Erectile Function (IIEF). Answers to qualitative questions are rated from 0 to 5, with a higher number indicating better erectile function, and totaled for a score which categorizes severity of erectile dysfunction. Total scores range from 5 to 25, with a lower score indicating more severe erectile dysfunction.
Time Frame: Assessed at Baseline, 4 Weeks, 8 Weeks, and 20 Weeks; change from Baseline at week 20 reported.
Measure: Mean (Full Range); unit: Score on a scale
Arm/Group | Percutaneous Epidural Stimulation | Transcutaneous Epidural Stimulation
Number analyzed (Participants) | 3 | 2
Score on a scale | -23.3 [-35 to -11] | -1.5 [-2 to -1]

10. Primary Outcome: Female Patient-reported Sexual Function
Description: Measurement of change in sexual function using the Female Sexual Function Index (FSFI). Answers to qualitative questions are rated from 0 to 5, with a higher number indicating better sexual function, and totaled for a score which categorizes severity of sexual dysfunction.
Time Frame: Assessed at Baseline, 4 Weeks, 8 Weeks, and 20 Weeks; change from Baseline at week 20 reported.
Population: No female participants were enrolled.
Arm/Group | Percutaneous Epidural Stimulation | Transcutaneous Epidural Stimulation
Number analyzed (Participants) | 0 | 0

11. Primary Outcome: Spasticity
Description: Change in measurements of spasticity using the Spinal Cord Injury Spasticity Evaluation Tool (SCI-SET). Answers to qualitative questions are rated from -3 to +3, with a higher positive number indicating more helpful symptoms, and a lower negative number indicating more problematic symptoms. Questions may also be answered as not applicable (N/A), which do not generate a score. Scores are totaled for a score which categorizes the overall positive or negative impact of a subject's spasticity symptoms. Total score can range from -105 (negative impact) to +105 (positive impact), and the score is averaged by total positive or negative score divided by the number of applicable answers.
Time Frame: Assessed at Baseline, 4 Weeks, 8 Weeks, and 20 Weeks; change from Baseline at week 20 reported.
Measure: Median (Full Range); unit: Score on a scale
Arm/Group | Percutaneous Epidural Stimulation | Transcutaneous Epidural Stimulation
Number analyzed (Participants) | 3 | 2
Score on a scale | 0.057 [-0.033 to 0.090] | 0.088 [-0.207 to 0.383]

12. Primary Outcome: Neurostimulation User Experience
Description: Rating of the subject's perception of individual aspects of spinal stimulation using the User Experience Questionnaire (UEQ), a survey including 26 descriptive terms and their antonyms. A scoring scale ranging from 1 to 7 determines how closely the subject feels the term or its antonym applies to the intervention, with lower numbers indicating agreement with the term, and higher numbers indicating agreement with the antonym. The terms and antonyms describe a positive and negative perception of each item.
  Subscales grouping terms into like categories average scores into a 7 point range from -3 to +3, with negative averages associated with negative perceptions, and positive averages associated with positive perceptions.
Time Frame: End of intervention, an average of 4 weeks
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Percutaneous Epidural Stimulation | Transcutaneous Epidural Stimulation
Number analyzed (Participants) | 3 | 2
Score on a scale
  Attractiveness | 3 (0) | 2.5 (0)
  Perspicuity | 1.5 (0.707) | 1.917 (0.382)
  Efficiency | 2.583 (0.382) | 2 (0.354)
  Dependability | 2.083 (0.520) | 1.75 (0.354)
  Stimulation | 2.917 (0.144) | 2 (0.354)
  Novelty | 2.583 (0.382) | 1.75 (1.414)

13. Primary Outcome: Overground Ambulation [as Appropriate to the Subject]
Description: Measurement of changes in overground mobility as measured by the Modified 6 Minute Walk Test. Trainers will assess the distance in meters which the subject can cover in 6 minutes, with a greater distance characterizing better overground mobility.
Time Frame: Baseline, 4 Weeks, 8 Weeks, and 20 Weeks
Population: No Transcutaneous Epidural Stimulation arm participants were ambulatory.
Measure: Number; unit: meters
Arm/Group | Percutaneous Epidural Stimulation | Transcutaneous Epidural Stimulation
Number analyzed (Participants) | 1 | 0
meters
  Pre-intervention to post-intervention | 9.2 |
  Pre-intervention to 8 weeks post intervention | 16.5 |
  Pre-intervention to 20 weeks post intervention | 16.5 |

14. Primary Outcome: Trunk Stability
Description: Changes in trunk stability based on stable forward reach measured in centimeters, with a greater distance of forward reach characterizing greater trunk stability. Specifically, change in forward reach at the end of the study when comparing stimulation assisted reach and non-stimulation assisted reach.
Time Frame: Beginning of intervention to end of intervention, an average of 17 days, 8 weeks post beginning of intervention, 20 weeks post beginning of intervention; change from beginning of intervention at week 20 reported.
Measure: Mean (Standard Deviation); unit: centimeters
Arm/Group | Percutaneous Epidural Stimulation | Transcutaneous Epidural Stimulation
Number analyzed (Participants) | 3 | 2
centimeters
  Non-stimulation assisted reach | 14.933333 (9.3972809) | 3 (3)
  Stimulation assisted reach | 34.933333 (14.115319) | 21.5 (11)

15. Primary Outcome: Neurostimulator Lead Location and Migration [Epidural Group Only]
Description: Evaluation of current array location via CT.
Time Frame: Pre-intervention and 4 weeks post-intervention
Population: Analysis applies only to percutaneous group participants.
Measure: Median (Full Range); unit: millimeters
Arm/Group | Percutaneous Epidural Stimulation | Transcutaneous Epidural Stimulation
Number analyzed (Participants) | 3 | 0
millimeters | -5.35862 [-8.48728 to -2.48357] |

16. Primary Outcome: Bladder Function Testing
Description: Change in measurements of bladder function (end fill detrusor value) utilizing a urodynamic test consisting of a filling phase and a voiding phase cystometrogram along with perineal patch muscle electromyography.
Time Frame: Beginning of study, prior to initiating intervention; End of 4 weeks of intervention.
Measure: Mean (Standard Deviation); unit: cm H2O
Arm/Group | Percutaneous Epidural Stimulation | Transcutaneous Epidural Stimulation
Number analyzed (Participants) | 3 | 2
cm H2O
  Pre-intervention | 21 (15.769168) | 10.5 (5.5)
  Post-intervention | 54.666667 (32.148959) | 15 (15)

ADVERSE EVENTS:
Time Frame: Adverse events were assessed over the course of approximately 20 weeks.
Arm/Group | Percutaneous Epidural Stimulation | Transcutaneous Epidural Stimulation
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/3 | 1/3
Other Adverse Events (participants affected / at risk) | 1/3 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Percutaneous Epidural Stimulation (N=3) | Transcutaneous Epidural Stimulation (N=3)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1) — Subject experienced mild hydronephrosis secondary to obstructing renal calculus, with hospitalization and subsequent ureteral stent placement, and calculus and stent removal.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Percutaneous Epidural Stimulation (N=3) | Transcutaneous Epidural Stimulation (N=3)
Petechiae (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 1 (2) | 0 (0)
Serosanguinous drainage (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Urinary tract infection (Renal and urinary disorders) | 1 (1) | 2 (3)
Urethral irritation post urodynamics study (Renal and urinary disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 2 (2)
Low back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1)
COVID-19 infection (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Bowel incontinence (Gastrointestinal disorders) | 0 (0) | 2 (2)
Skin irritation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Autonomic dysreflexia (Nervous system disorders) | 0 (0) | 1 (3)
Hemorrhoids (Vascular disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-11-07): https://cdn.clinicaltrials.gov/large-docs/54/NCT05095454/Prot_SAP_000.pdf
  • Informed Consent Form (2022-12-14): https://cdn.clinicaltrials.gov/large-docs/54/NCT05095454/ICF_001.pdf